CLINICAL TRIAL: NCT07118319
Title: A Phase I Study to Assess the Safety, Tolerability and Preliminary Efficacy of Human Allogeneic Induced Pluripotent Stem Cells (iPSCs) -Derived Motor Neuron Progenitor Cells (XS228CN) in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: The Safety, Tolerability and Preliminary Efficacy of Derived Motor Neuron Progenitor Cells (XS228CN) in Subjects With Amyotrophic Lateral Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: XellSmart Bio-Pharmaceutical (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XS228-Allo-ALS-CN1/2-P01; 2025LP01221 (Registry Identifier: China Center for Drug Evaluation (CDE), NMPA)
Record Dates: First submitted 2025-07-24; First posted 2025-08-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5.0×10^7 cells/person/dose (Experimental): intrathecal injection
  Interventions: Drug: Human Allogeneic Induced Pluripotent Stem Cells (iPSCs) -Derived Motor Neuron Progenitor Cells (XS228CN)
- 1.0×10^8 cells/person/dose (Experimental): intrathecal injection
  Interventions: Drug: Human Allogeneic Induced Pluripotent Stem Cells (iPSCs) -Derived Motor Neuron Progenitor Cells (XS228CN)

INTERVENTIONS:
Drug: Human Allogeneic Induced Pluripotent Stem Cells (iPSCs) -Derived Motor Neuron Progenitor Cells (XS228CN) — Injection, once, 6 months
Drug: Human Allogeneic Induced Pluripotent Stem Cells (iPSCs) -Derived Motor Neuron Progenitor Cells (XS228CN) — Injection, every two weeks for four doses, 6 months

SUMMARY:
A Phase I Study to Assess the Safety, Tolerability and Preliminary Efficacy of Derived Motor Neuron Progenitor Cells (XS228CN) in Subjects with Amyotrophic Lateral Sclerosis

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age (inclusive of 18 and 75 years), regardless of gender;
2. Diagnosed of definite or probable ALS according to the revised EI Escorial criteria;
3. Respiratory function FVC at baseline was ≥70% of the predicted value (FVC%);
4. Patients with birth-potential (both male and female) must agree to use effective non-drug contraceptive measures from the time of signing the informed consent until 6 months after the conclusion of the trial;
5. Volunteer to participate in the clinical study, understand and sign the informed consent form.

Exclusion Criteria:

1. Subject has signs and symptoms of neuromuscular weakness, and other causes of muscle weakness cannot be ruled out;
2. Baseline body mass index (BMI) < 18.5 kg/m²;
3. Primary lateral sclerosis presenting only with upper motor neuron symptoms;
4. Significant psychiatric disorders that the investigator assesses may affect evaluation;
5. Diseases causing neurological or muscular dysfunction, such as metabolic muscle diseases or myasthenia gravis;
6. Diagnosed autoimmune diseases with uncontrolled severe arthritis or other conditions (e.g., lameness) that the investigator assesses may affect evaluation;
7. Acute active infections requiring antibiotics, antivirals, or antifungals that occurred within the 2 weeks prior to screening and are not controlled;
8. Subject diagnosed with active pulmonary tuberculosis or treated for suspected tuberculosis;
9. Diagnosed severe pulmonary diseases that the investigator assesses may affect evaluation;
10. Poorly controlled hypertension;
11. Previous or detected cardiac abnormalities;
12. A history of cirrhosis, chronic hepatitis, or liver function at screening;
13. A history of chronic kidney disease;
14. Previous history of bleeding, abnormal clotting, or being treated with anticoagulation;
15. Active hepatitis B, active hepatitis C, human immunodeficiency virus (HIV) antibody or treponema pallidum antibody positive at screening;
16. History of severe trauma or surgery and may affect the assessment judged by investigator;
17. Subjects with contraindications to lumbar puncture, including menifestations of injection site infection or high intracranial pressure.
18. Those who have had a malignant tumor within 5 years prior to screening or are undergoing antitumor therapy;
19. Have participated in other clinical trials within 3 months prior to screening;
20. Pregnant or breastfeeding women;
21. Subject who is judged by the investigator to be unsuitable for the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of XS228CN-related adverse events (AEs) and serious adverse events (SAEs) within 28 days after the last administration in ALS patients | within 28 days after the last administration

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes